CLINICAL TRIAL: NCT06351241
Title: Hemodynamic Effects of Steep Trendelenburg Position and Pneumoperitoneum in Urologic Robotic Surgery: a Prospective Study
Brief Title: Hemodynamic Effects of Steep Trendelenburg Position and Pneumoperitoneum
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Nursen Karaca, Principal Investigator, Ege University
Other Study IDs: E.222840/280
Record Dates: First submitted 2024-03-18; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Perfusion Index; Pleth Variability Index
Keywords: Perfusion index; Pleth variability index; Robotic surgery; Pneumoperitoneum; Steep trendelenburg position
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
BACKGROUND: The steep Trendelenburg position and pneumoperitoneum are used to improve surgical visibility in robot-assisted laparoscopic radical prostatectomy (RALRP). However, these procedures can lead to hemodynamic changes. This study aimed to investigate the effects of these interventions on the perfusion index (PI) and the Pleth variability index (PVI) in patients undergoing RALRP under general anesthesia.

METHODS: Fifty-three patients scheduled for RALRP underwent standard monitoring; PI and PVI values were monitored using a finger probe. PI, PVI, hemodynamic and respiratory parameters, and intraabdominal pressure were recorded before and after anesthesia induction, after adopting the Trendelenburg position, after pneumoperitoneum, after pneumoperitoneum and the Trendelenburg position, at 15 min, 30 min, in the supine position, after carbon dioxide (CO2) desufflation, and after extubation.

DETAILED DESCRIPTION:
Introduction Robot-assisted laparoscopic radical prostatectomy (RYLRP) is currently the most frequently performed surgical procedure using the Da Vinci Robotic System. In this procedure, the steep Trendelenburg position (30° - 45° head down) and pneumoperitoneum (insufflation of the intraabdominal space with CO2) are used to enhance surgical visibility in the retroperitoneal area. However, the patient position and pneumoperitoneum used in robotic surgery can lead to fluctuations in hemodynamic parameters resulting from physiological changes in the cardiovascular and respiratory systems. Consequently, proper hemodynamic monitoring and optimal fluid management can reduce the risk of complications and improve outcomes in patients.

Perfusion index (PI) is a hemodynamic parameter calculated by looking at the absorption of infrared light by pulse oximetry to evaluate continuous tissue perfusion for a specific time interval. In contrast, the Pleth variability index (PVI), a dynamic variable used for regulating fluid management, is computed based on changes in PI caused by ventilation over at least one respiratory cycle. Both parameters are key non-invasive methods for hemodynamic monitoring during patient follow-up as they provide accurate information about tissue perfusion. However, only a few studies have evaluated the effects of patient position and pneumoperitoneum on PI and PVI in laparoscopic surgeries. Therefore, this study aimed to prospectively investigate the effects of the steep Trendelenburg position and pneumoperitoneum on PVI and PI in patients scheduled for RYLRP under general anesthesia.

Materials and methods This prospective observational study was approved by the Ege University Faculty of Medicine Clinical Research Ethics Committee (approval number: E222840/280; dated July 7, 2021). Patients belonging to ASA classes I-II, aged between 25 and 80 years, and scheduled for elective RYLRP under general anesthesia were included in the study. Patients deemed suitable for the study were explained about the study, and written voluntary informed consent for participation was obtained. Two patients were eventually dropped from the study because of conversion to open surgery. Additionally, patients with an ASA score above III, those unsuitable for robotic surgery, and those who developed hemodynamic instability or respiratory complications during the intraoperative period were excluded.

Preanesthetic evaluations of the patients were performed at least 24 hour before the operation. Preoperative data, including age, weight, height, body mass index, ASA classification, and additional medical history, were recorded for each patient.

After being admitted to the operating room, standard monitoring (electrocardiogram, non-invasive blood pressure, peripheral oxygen saturation) was performed. In addition, non-invasive hemoglobin, PI, and PVI monitoring were conducted using a finger probe (Masimo Radikal 7, Masimo Corp., Irvine, CA, USA) which was placed on the fourth digit of the hand without the non-invasive blood pressure cuff. A 16-G or 18-G intravenous (IV) cannula was inserted, and an Isolyte-S infusion was initiated.

After 3 min of pre-oxygenation with 100% O2, standard anesthesia induction (using 0.5 mg atropine, 1 mg/kg lidocaine, 2 - 3 mg/kg propofol, 1-3 µg/kg fentanyl, and 0.6 mg/kg rocuronium bromide) was performed. Following adequate mask ventilation, the patients were intubated with an endotracheal tube with an internal diameter of 7.5 - 8.5 mm. The endotracheal tube placement was verified by confirming equal ventilation in both lungs and observing the end-tidal carbon dioxide (ETCO2) waveform in the capnograph. Patients were then placed on volume-controlled mechanical ventilation with a tidal volume of 6-8 mL/kg and ETCO2 maintained at 35 - 40 mmHg. Invasive arterial blood pressure measurements were performed via radial artery cannulation throughout the operation. Anesthesia maintenance included a mixture of 50 % O2 and air with 2 % MAC sevoflurane (Sevoflurane Liquid 250 ml®, Abbott, UK) and remifentanil infusion.

After anesthesia induction and intubation, the patients were placed in a 45° steep Trendelenburg position. Five minutes after positioning, hemodynamic and respiratory parameters were recorded, and the patients were returned to the supine position. After returning to the supine position, pneumoperitoneum was established with CO2, and hemodynamic and respiratory parameters were recorded again 5 min later.

Measurements were taken at the following time points: before anesthesia induction (T0), 5 min after induction (T1), 5 min after the steep Trendelenburg position was applied (T2), 5 min after establishing pneumoperitoneum (T3), 5 min (T4), 15 min (T5) and 30 min (T6) after pneumoperitoneum and the steep Trendelenburg position were applied together, upon returning to the supine position (T7), after CO2 desufflation (T8), and after extubation (T9). The following parameters were recorded: hemodynamic parameters (systolic blood pressure, diastolic blood pressure, mean arterial pressure, heart rate, PI, and PDI), respiratory parameters (tidal volume, respiratory rate, peak airway pressure, mean airway pressure, PEEP, ETCO2, oxygen saturation (SpO2), and compliance), intraabdominal pressure, non-invasive hemoglobin, and body temperature. At the end of the surgery, the operation time, anesthesia time, pneumoperitoneum duration, intraoperative fluid volume administered, urine output, and intraoperative bleeding amount were recorded (Figure 1).

The data so collected were analyzed using IBM SPSS (version 23.0; IBM Corp., Armonk, NY). Frequency and percentage were computed for categorical data, whereas mean, standard deviation (SD), median, and range were presented as descriptive values for continuous data. Friedman's two-way analysis of variance by rank was employed to assess the differences between dependent measurements at different time points. A p-value of 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients belonging to ASA classes I-II
* Aged between 25 and 80 years
* Elective robot-assisted laparoscopic radical prostatectomy under general anesthesia

Exclusion Criteria:

* conversion to open surgery
* patients with an ASA score above III
* unsuitable for robotic surgery
* who developed hemodynamic instability or respiratory complications during the intraoperative period

Ages: 25 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients belonging to ASA classes I-II, aged between 25 and 80 years, and scheduled for elective robot-assisted laparoscopic radical prostatectomy under general anesthesia were included in the study. Patients deemed suitable for the study were explained about the study, and written voluntary informed consent for participation was obtained.
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Hemodynamic effects of steep trendelenburg position and pneumoperitoneum in urologic robotic surgery | 1 year
  Can steep trendelenburg position and pneumoperitoneum cause hemodynamic changes in urologic robotic surgery? Hemodynamic measurements were taken at specific time points during the operation. The following hemodinamic parameters, Perfusion index (PI) and Pleth variability index, were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Işık Alper, Study Director — Ege University
Locations (1):
- Nursen Karaca, Bornova, İzmir, Turkey (Türkiye)